CLINICAL TRIAL: NCT01806961
Title: Observational (Non-interventional), Follow-up Trial Assessing Long-term Local Tolerability and Efficacy (Recurrence Rate) of Resiquimod Gel in Patients Treated for Actinic Keratosis.
Brief Title: Observational Trial Tolerability and Efficacy of Resiquimod Gel in Patients Treated for Actinic Keratosis.
Status: Terminated | Type: Observational
Why Stopped: sponsor decision
Sponsor: Spirig Pharma Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: SP848-AKEx-1209
Record Dates: First submitted 2013-03-06; First posted 2013-03-07 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-05

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- clearance at end of trial SP848-AK-1101: no trial medication during this follow-up trial

SUMMARY:
Determine the recurrence rate of actinic keratosis (AK) lesions in patients with complete clinical clearance at the end of the previous trial SP848-AK-1101 at 6 and 12 months of follow-up.

DETAILED DESCRIPTION:
Efficacy Evaluation:

• Primarily based on clinical inspection of the former 25 cm2 treatment area and count of the AK-lesions.

Safety Evaluation:

* Evaluation of adverse events (AEs) and serious adverse events (SAEs)
* Evaluation of newly occurred dermal adverse events (AEs) and serious adverse events (SAEs) in the previous treatment area at 6 months and 12 months of follow-up (local tolerability).
* Follow-up of unresolved adverse and serious adverse events that occurred in the previous trial SP848-AK-1101.
* Follow-up of unresolved abnormal laboratory values that occurred in the previous trial SP848-AK-1101.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Participation in the previous clinical trial SP848-AK-1101.
* Patient with complete clinical clearance (i.e. no previously existing AK-lesion present) at the end of the trial SP848-AK-1101 or Non-Responder who withdrew from the trial prematurely.

Exclusion Criteria:

* Evidence of unstable or uncontrolled clinically significant medical conditions as determined by the investigator (e.g., cardiovascular, immunological, hematologic, hepatic, neurologic, renal, endocrine, collagen-vascular, infectious, gastrointestinal abnormalities or diseases).
* Evidence of systemic cancer.
* Dermatological disease or condition in the former treatment or surrounding area that might impair trial assessments (e.g., rosacea, atopic dermatitis, eczema) as assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with complete clinical clearance (i.e. no previously existing AK-lesion present) at the end of the trial SP848-AK-1101 or Non- Responder who withdrew from the trial prematurely.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars E French, MD, Principal Investigator — University Clinic of Dermatology, Zurich
Locations (9):
- Germany (5):
  - Hauttumorcentrum Charité (HTCC), Berlin
  - Medizinisches Zentrum Bonn - Friedensplatz, Bonn
  - Hautzentrum, Düsseldorf
  - Johannes Wesling Klinikum Minden, Minden
  - KLINIKUM VEST GmbH Knappschaftskrankenhaus, Recklinghausen
- Switzerland (4):
  - Universitätsspital Basel, Basel
  - Inselspital, Bern
  - Kantonsspital St.Gallen, Sankt Gallen
  - Universitaetsspital Zurich, Zurich

RESULTS

PARTICIPANT FLOW:
Groups:
- SP848-AK-1101: Patients from SP848-AK-1101 trial
Period: Overall Study
Arm/Group | SP848-AK-1101
Started | 16
Completed | 0
Not Completed | 16
Not completed — sponsor decision | 16

BASELINE CHARACTERISTICS:
Arm/Group | Clearance at End of Trial SP848-AK-1101
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 73 [53 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Determine the Recurrence Rate of AK-lesions
Description: Number of patients with persistent complete clearance at 6 and 12 months follow-up. Recurrence rate is to be determined at the same treatment area where the investigational medicinal products were administered in the previous trial.
Time Frame: at 6 and 12 months
Population: No subject was analysed due to premature study termination (sponsor's decision) therefore no data was available for analysis
Groups:
- Group 1: Patients from SP848-AK-1101 trial
Arm/Group | Group 1
Number analyzed (Participants) | 0

2. Secondary Outcome: Follow-up of AK-lesions (Existing Lesions, New Lesions, Changes)
Description: clinical examination
Time Frame: at 6 and 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Number of Newly Occurred Dermal Adverse and Serious Adverse Events on the Previous Treatment Area
Description: recording of adverse events
Time Frame: at 6 and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 6/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=16)
Basal cell carcinome lower back (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=16)
unspecific inflammation crus helicis left arm (General disorders) | 1 (1)
common cold (Infections and infestations) | 1 (1)
wart (Skin and subcutaneous tissue disorders) | 2 (2)
oesophageal acid reflux (Gastrointestinal disorders) | 1 (1)
sinusitis (Infections and infestations) | 1 (1)
hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1)
carotid stenosis (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
No efficacy analysis was carried out since due to premature study termination (upon Sponsor's decision) no data was available for analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the PI and the Sponsor that restricts the PI's rights to discuss or publish trial results after the trial is completed.

Investigator is granted a right to publish and present Trial Results together with other investigators of Trial and to be referred to in publications containing such results. However, PI shall not publish or present Results unless Investigator has submitted to Spirig a draft of the intented publication or presentation for review and approval.